CLINICAL TRIAL: NCT02195531
Title: BIG4 - CPAP Educational Materials and Usage Feedback to Promote CPAP Adherence
Brief Title: CPAP (Continuous Positive Airway Pressure) Study Educational Materials and Usage Feedback to Promote CPAP Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Respironics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PGI-BIG4-1331-MS
Record Dates: First submitted 2014-07-14; First posted 2014-07-21 (Estimated); Results first posted 2019-04-05 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-01

CONDITIONS: Adherence
Keywords: Adherence
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment (Active Comparator): Participants will receive education and feedback tailored to the psychological profile of the receiving participant.
  Interventions: Behavioral: Education and feedback
- Control Group (Active Comparator): Participants will receive education inconsistent with their profile.
  Interventions: Behavioral: Education and feedback
- Standard of care (No Intervention): Participants will not receive education or feedback.

INTERVENTIONS:
Behavioral: Education and feedback — The education leaflets are information concerning Obstructive Sleep Apna (OSA) and CPAP treatment. The feedback reports are CPAP usage patterns.
  Other Names: Education; Motivational Enhancement technique
  Arms: Control Group; Treatment

SUMMARY:
The study hypothesis: in groups receiving tailored education and feedback in a style that matches their psychological profile, will show a higher CPAP adherence rates than groups receiving mismatched tailored education / feedback, and groups that receive no tailored education and feedback (standard of care).

DETAILED DESCRIPTION:
Three group, randomized, controlled clinical trial assessing the extent to which tailoring a CPAP intervention entailing education and feedback to the psychological profile of new CPAP users can enhance the impact of the intervention in terms of adherence-related behavior.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, ages 21-80 years
* Prescribed to start CPAP treatment and diagnosed with mild to severe OSA.
* Recently (within study period) diagnosed with Mild to Severe OSA defined as an Apnea-Hypopnea Index of equal to or greater than 10 events per hour of sleep.
* CPAP treatment naïve

Exclusion Criteria:

* Inability to provide informed consent
* Presence of a comorbid condition that may potentially complicate CPAP adherence, such as:

  * Unstable depressive disorder
  * Unstable anxiety disorder
  * Dementia
  * Unable to understand study information
  * Obesity Hypoventilation Syndrome
  * Central Sleep Apnea or Complex Sleep Apnea
  * Facial musculoskeletal disorder

    * Unwillingness or inability to use CPAP therapy
    * Unable to return for follow up appointment
    * Use of supplemental oxygen

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2014-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bogan, MD, Principal Investigator — SleepMed of South Carolina
Locations (6):
- United States (6):
  - Pulmonary Associates, Glendale, Arizona
  - Arkansas Center for Sleep Medicine, Little Rock, Arkansas
  - NeuroTrials, Inc., Atlanta, Georgia
  - SleepMed of Central Georgia, Macon, Georgia
  - SleepMed of Philadelphia, Philadelphia, Pennsylvania
  - SleepMed of South Carolina, Columbia, South Carolina

REFERENCES:
- [Derived] Lacroix J, Tatousek J, Den Teuling N, Visser T, Wells C, Wylie P, Rosenberg R, Bogan R. Effectiveness of an Intervention Providing Digitally Generated Personalized Feedback and Education on Adherence to Continuous Positive Airway Pressure: Randomized Controlled Trial. J Med Internet Res. 2023 May 22;25:e40193. doi: 10.2196/40193. PMID 37213195

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group: Participants will receive education and feedback tailored to the psychological profile of the receiving participant.
  Education and feedback: The education leaflets are information concerning OSA and CPAP treatment. The feedback reports are CPAP usage patterns.
- Control Group: Participants will receive education inconsistent with their profile.
  Education and feedback: The education leaflets are information concerning OSA and CPAP treatment. The feedback reports are CPAP usage patterns.
Period: Overall Study
Arm/Group | Standard of Care | Treatment Group | Control Group
Started | 64 | 49 | 56
Completed | 63 | 48 | 55
Not Completed | 1 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Treatment: Participants will receive education and feedback tailored to the psychological profile of the receiving participant.
  Education and feedback: The education leaflets are information concerning OSA and CPAP treatment. The feedback reports are CPAP usage patterns.
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Treatment | Control Group | Total
Number analyzed (Participants) | 63 | 48 | 55 | 166
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.0 (12.5) | 50.5 (10.9) | 53.3 (12.8) | 50.5 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 14 | 17 | 54
  Male | 40 | 34 | 38 | 112
Region of Enrollment [Number; unit: participants]
  United States | 63 | 48 | 55 | 166
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 34.5 (8.2) | 32.8 (5.6) | 33.6 (6.5) | 33.7 (7.0)
Apnea-Hyopnea Index [Mean (Standard Deviation); unit: events/hour] — The apnea-hypopnea index (AHI) is the combined average number of apneas and hypopneas that occur per hour of sleep
  events/hour | 32.7 (17.9) | 27.1 (16.1) | 28.2 (16.2) | 29.6 (17.0)
Epworth Sleepiness Scale [Mean (Standard Deviation); unit: units on a scale] — The Epworth Sleepiness Scale is an 8 item questionnaire that measures the general level of daytime sleepiness. Participants were asked what the chance is they would doze off or fall asleep during different routine daytime situations. The survey answers questions on a scale of 0 to 3- 0 being no chance and 3 being a high chance of dozing. The lowest score possible is a 0 and the highest score possible is a 24.
  units on a scale | 11.1 (5.6) | 10.4 (5.3) | 11.2 (5.6) | 10.9 (5.5)

OUTCOME MEASURES:

1. Primary Outcome: Nightly Adherence
Description: Average usage hours per night
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Treatment | Control Group | Standard of Care
Number analyzed (Participants) | 48 | 55 | 63
hours
  Week 1 | 4.83 (3.04) | 5.82 (3.08) | 4.82 (2.90)
  Month 1 | 4.60 (3.09) | 4.96 (3.09) | 4.19 (3.05)
  Month 2 | 4.32 (3.10) | 4.94 (3.08) | 3.60 (3.23)
  Month 3 | 4.16 (3.18) | 4.63 (3.27) | 3.25 (3.27)

2. Primary Outcome: Adherence
Description: Average usage days per week.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: days per week
Arm/Group | Treatment | Control Group | Standard of Care
Number analyzed (Participants) | 48 | 55 | 63
days per week | 5.5 (2.1) | 5.8 (1.7) | 4.9 (2.5)

3. Secondary Outcome: Participant's Feedback on Educational Pamphlets - Expectations Scale
Description: Explore the difference in efficacy of the educational and feedback materials tailored to the specific psychological profiles.
  Participants answered 3 questions about the expected effectiveness of CPAP. These questions were on a scale of 0 to 5, 0 being not effective at all and 5 being extremely effective.
  The average response for each questions was analyzed.
Time Frame: 3 months
Population: As the study progressed participants withdrew or were withdrawn from the study. Or they did not complete the assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment | Control Group | Standard of Care
Number analyzed (Participants) | 48 | 55 | 63
units on a scale
  Screening | 4.42 (0.63) | 4.39 (0.80) | 4.33 (0.72)
  Month 1: number analyzed (Participants) | 45 | 51 | 50
  Month 1 | 4.10 (0.85) | 4.01 (1.01) | 4.07 (0.65)
  Month 2: number analyzed (Participants) | 43 | 53 | 61
  Month 2 | 4.43 (0.70) | 4.26 (0.85) | 3.97 (0.88)
  Month 3: number analyzed (Participants) | 44 | 52 | 59
  Month 3 | 4.33 (0.73) | 4.30 (0.79) | 3.99 (1.03)

4. Secondary Outcome: Participant's Feedback on Educational Pamphlets - Importance Scale
Description: Explore the difference in efficacy of the educational and feedback materials tailored to the specific psychological profiles.
  Participants answered one questions about the importance of CPAP. This was was on a scale of 0 to 5, 0 being not important at all and 5 extremely important.
Time Frame: 3 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment | Control Group | Standard of Care
Number analyzed (Participants) | 48 | 55 | 63
units on a scale
  Screening | 4.69 (0.59) | 4.58 (0.71) | 4.65 (0.65)
  Month 1: number analyzed (Participants) | 45 | 51 | 50
  Month 1 | 4.53 (0.87) | 4.63 (0.72) | 4.62 (0.67)
  Month 2: number analyzed (Participants) | 43 | 53 | 61
  Month 2 | 4.65 (0.65) | 4.66 (0.71) | 4.36 (0.82)
  Month 3: number analyzed (Participants) | 44 | 52 | 59
  Month 3 | 4.86 (0.41) | 4.73 (0.60) | 4.31 (0.99)

5. Secondary Outcome: Participant's Feedback on Educational Pamphlets - Self-Efficacy Scale
Description: Explore the difference in efficacy of the educational and feedback materials tailored to the specific psychological profiles.
  Participants answered 5 questions regarding self-efficacy of use of CPAP. This was on a scale of 0 to 5, 0 being disagree completely and 5 being completely agree.
  The average of each question was analyzed.
Time Frame: 3 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment | Control Group | Standard of Care
Number analyzed (Participants) | 48 | 55 | 63
units on a scale
  Screening | 4.49 (0.53) | 4.20 (0.84) | 4.29 (0.73)
  Month 1: number analyzed (Participants) | 45 | 51 | 50
  Month 1 | 4.26 (0.79) | 4.14 (0.86) | 4.07 (0.85)
  Month 2: number analyzed (Participants) | 43 | 53 | 61
  Month 2 | 4.29 (0.76) | 4.42 (0.81) | 4.14 (1.00)
  Month 3: number analyzed (Participants) | 44 | 52 | 59
  Month 3 | 4.28 (0.98) | 4.30 (0.89) | 4.04 (1.08)

6. Secondary Outcome: Participant's Feedback on Educational Pamphlets - Motiviation
Description: Explore the difference in efficacy of the educational and feedback materials tailored to the specific psychological profiles.
  Participants were asked about there motivation to use CPAP with two questions. These questions were on a scale of 0 to 10, 0 being not at all, 5 being somewhat, and 10 very much.
  The average of the questions were analyzed.
Time Frame: 3 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment | Control Group | Standard of Care
Number analyzed (Participants) | 48 | 55 | 63
units on a scale
  Screening | 9.59 (0.56) | 9.32 (1.14) | 9.21 (1.40)
  Month 1: number analyzed (Participants) | 45 | 51 | 50
  Month 1 | 9.10 (1.35) | 8.82 (1.75) | 8.85 (1.47)
  Month 2: number analyzed (Participants) | 43 | 53 | 61
  Month 2 | 9.38 (0.97) | 9.25 (1.59) | 8.97 (1.57)
  Month 3: number analyzed (Participants) | 44 | 52 | 59
  Month 3 | 9.11 (1.23) | 8.98 (1.81) | 8.57 (1.83)

7. Secondary Outcome: Participant's Feedback on Educational Pamphlets - Leaflet Assessment
Description: Explore the difference in efficacy of the educational and feedback materials tailored to the specific psychological profiles.
  Participants that received the leaflet were asked 15 questions regarding it. The questions were on a scale of 0 to 5, 0 being strongly disagree and 5 being strongly agree.
  The average of the scores were calculated and analyzed monthly.
Time Frame: 2 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment | Control Group
Number analyzed (Participants) | 48 | 55
units on a scale
  Screening | 4.12 (0.46) | 4.04 (0.63)
  Month 1: number analyzed (Participants) | 45 | 51
  Month 1 | 3.94 (0.58) | 3.95 (0.72)
  Month 2: number analyzed (Participants) | 43 | 53
  Month 2 | 4.07 (0.74) | 3.99 (0.73)

ADVERSE EVENTS:
Time Frame: All non-serious and serious adverse events were collected over the 3 month period
Arm/Group | Treatment | Control Group | Standard of Care
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/55 | 0/63
Other Adverse Events (participants affected / at risk) | 0/48 | 0/55 | 0/63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No